CLINICAL TRIAL: NCT07320378
Title: Clinical Study on the Safety and Efficacy of Tendon Stem Progenitor Cells Therapy for Rotator Cuff Tears
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-1814
Record Dates: First submitted 2025-11-24; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tendinopathy

STUDY DESIGN:
Intervention Model Description: In the Phase I of this clinical study, we will design a dose-escalation clinical study to evaluate the maximum tolerated dose (MTD) and safety of tendon stem/progenitor cell (TSPC)-enhanced rotator cuff repair. In the Phase II of the study, we will design a randomized controlled trial (RCT) to assess the efficacy of TSPC-enhanced rotator cuff repair.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In phase II clinical trial, blinding will be applied to the participants, those measuring the intervention effects, and the statistician responsible for the analysis. The operating surgeons will not be blinded. Sequentially numbered, sealed opaque envelopes containing group allocation information will be provided to the operating surgeons. Group allocation concealment will be ensured through the use of a central automated randomization system, and security measures will be implemented to prevent those blinded from accessing or influencing the allocation data. Objective measurements of rotator cuff structural changes and pain will be performed by trained assessors unaware of the group assignments. The statistician conducting the statistical analysis will also remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery group (Active Comparator): All procedures were performed under general anesthesia, including subacromial decompression, acromioplasty, and rotator cuff repair using a double-row suture bridge technique.
  Interventions: Procedure: Conventional rotator cuff repair.
- TSPCs enhanced group (Experimental): For patients in the TSPCs group, after removing the arthroscopic fluid, TSPCs mixed with fibrin glue were applied to the tendon-bone junction and repaired tendon surface under arthroscopic guidance.
  Interventions: Biological: Stem cell therapy; Procedure: Conventional rotator cuff repair.

INTERVENTIONS:
Biological: Stem cell therapy — For patients in the TSPCs group, after removing the arthroscopic fluid, the prepared TSPCs loaded on a scaffold were injected into the tendon - bone junction and over the repaired tendon using a spinal needle. Fibrin glue (Fibrin Sealant (Human), RAAS) served as the scaffold. The TSPCs suspension was first mixed with thrombin solution at a 3:1 ratio. Then, using the DUPLOJECT syringe support system (Fibrin Sealant (Human), RAAS), 2 ml of cell - thrombin suspension was combined with 2 ml of fibrinogen solution at a 1:1 ratio and applied to the repaired tendon surface. After extracting the arthroscopic fluid, this cell - thrombin - fibrinogen suspension was implanted under arthroscopic guidance. A probe was used to spread and adjust the fibrin glue to cover the repaired tendon - bone junction and tendon surface.
  Arms: TSPCs enhanced group
Procedure: Conventional rotator cuff repair. — All procedures were performed under general anesthesia. Patients were in a beach-chair position. After glenohumeral inspection, subacromial decompression was conducted, and acromioplasty was performed. After subacromial decompression, the upper surface of the greater tuberosity was abraded to create a bleeding cancellous bone bed. The footprint of the greater tuberosity was debrided. Rotator cuff repair was performed using a double-row suture bridge technique. For medial-row repair, a hole was punched in the greater tuberosity, and a bioabsorbable suture anchor was inserted. After the medial row was completed, the suture limbs were used to create suture bridges over the tendon. The lateral fixation points were placed, and the suture anchor was used for lateral-row fixation.

SUMMARY:
Tendon injury is one of the most common sports injuries, including local tissue degeneration at the tendon insertion site following inflammation caused by long-term joint movement, friction, or strain, as well as acute traumatic tendon tears and defects of varying degrees due to sports. It is a recognized therapeutic challenge in orthopedics and sports medicine. With the increase in people's physical activities and changes in work styles, tendon injuries have become increasingly prevalent, with at least 30 million tendon injury cases annually. Meanwhile, tendon injuries pose a significant threat to the careers of many elite athletes. Currently, clinical treatments for tendon injuries mainly remain at the stages of physical therapy, surgical suture, and transplantation. Although these treatments have certain effects, their efficacy is limited-primarily because adult tendons lack complete regenerative capacity. As a result, the quality of repaired tendons is far inferior to that of normal tendons, making them prone to tendon adhesion, poor structural and mechanical properties, and frequent re-rupture. Even autologous tendon transplantation can only achieve approximately 40% of the mechanical properties of normal tendons, accompanied by excessive scar tissue formation. Current therapeutic and tissue engineering approaches can only partially improve tendon repair quality, failing to induce complete tendon repair and regeneration. Therefore, exploring new and efficient strategies for the treatment and regeneration of tendon injuries is of great significance.

In recent years, cell therapy has brought new opportunities for improving the repair quality of soft tissues such as tendons. Tendon-derived cells are isolated and extracted from tendons. These cells not only possess stem cell characteristics similar to bone marrow mesenchymal stem cells but also highly express tendon-specific genes and proteins. Therefore, this study intends to first culture and expand tendon stem/progenitor cells (TSPCs) to form therapeutic agents, then apply TSPC-enhanced therapy intraoperatively to patients with rotator cuff tendinopathy, and evaluate its clinical safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years, regardless of gender;
2. Tear size classified as small (< 1 cm) or medium-sized (1 cm to 3 cm) according to the DeOrio and Cofield classification system;
3. Persistent shoulder pain or functional limitations despite at least 3 months of non-surgical treatment, with indications for arthroscopic rotator cuff repair;
4. Willing to sign the informed consent form and agree to participate in this study.

Exclusion Criteria:

1. Tear size classified as large (3 cm to 5 cm) or massive (> 5 cm) according to the DeOrio and Cofield classification, or Patte grade 3 tendon retraction;
2. Subscapularis tendon tear;
3. Complicated with anterior, posterior, or multidirectional shoulder joint instability;
4. Indications for repair of anterior or posterior labral injury;
5. Intra-articular injection of hyaluronic acid or corticosteroids within 3 months prior to the planned surgery;
6. Comorbidities that contraindicate arthroscopic shoulder surgery;
7. Local (shoulder, abdomen, buttocks) or systemic infection, osteomyelitis, or sepsis;
8. Diabetes mellitus, untreated thyroid disease, chronic kidney disease, or rheumatoid arthritis;
9. Immunodeficiency;
10. Chronic diseases involving coagulation or platelet aggregation, or severe coagulopathy;
11. Severe cardiovascular disease;
12. Stroke or acute cardiovascular event within 6 months prior to the planned surgery;
13. Weight loss > 30 kg for any reason within 12 months, or unexplained weight loss > 10 kg within 12 months;
14. Eating disorder or body dysmorphic disorder;
15. Alcohol/drug addiction or mental illness that may affect compliance with postoperative protocols;
16. Pregnant or lactating women;
17. Refusal to sign the informed consent form;
18. Other conditions deemed inappropriate by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Phase I：Incidence and severity of cell therapy related adverse events | In 12 weeks
  Incidence and severity of cell therapy related adverse events:Adverse events are defined as abnormal laboratory test results, symptoms or signs, and are graded using the Common Terminology Criteria for Adverse Events (CTCAE). Serious adverse events are defined as any grade 3 or 4 adverse events as specified in the CTCAE.
Phase II：Oxford Shoulder Score (OSS) | 24 weeks
  OSS is a patient-reported measure used to assess functional limitations following shoulder surgery. It consists of 12 items, each with five response categories, and scores can range from 0 (indicating the worst functional status) to 48 (indicating the best functional status).

SECONDARY OUTCOMES:
Constant-Murley Score (CMS) | Baseline,Post-op Week 12,Post-op Week 24,Post-op Week 48
  The CMS provides an assessment of both Individual parameters and clinical symptoms, which is sufficiently sensitive to reveal even small changes in function. The score consists of four domains : pain (15 points), activities of daily living (20 points), movement (40 points), and strength (25 points).
Range of Motion (ROM) | Baseline,Post-op Week 12,Post-op Week 24,Post-op Week 48
  The examiner passively moved the patient's upper extremity to the end range of flexion, abduction, internal rotation, and external rotation, ensuring movements were within the patient's comfort level. Internal and external rotation were measured at 90° of abduction.
Shoulder pain at rest | Baseline,Post-op Week 1,Post-op Week 4,Post-op Week 8,Post-op Week 12,Post-op Week 24,Post-op Week 48
  A Numerical Rating Scale from 0 to 10 with "0" representing no pain and "10" representing the worst pain imaginable in the preceding week.
Work status | Baseline,Post-op Week 12,Post-op Week 24,Post-op Week 48
  Normal duties, restricted duties/hours, not working.
Tendon Integrity Classification on MRI | Post-op Week 24, Post-op Week 48
  According to SUGAYA Classification.
Muscle wasting of rotator cuff on MRI | Baseline, Post-op Week 24, Post-op Week 48
  Measured using Goutallier classification (Stages 0-4).

IPD SHARING:
Plan to Share IPD: Undecided